CLINICAL TRIAL: NCT00884650
Title: Comparing the Effectiveness of an Anesthetic Continuous-infusion Device to Oral Analgesia in Orthopedic Postoperative Pain Control of Children With Cerebral Palsy
Brief Title: Managing Post-operative Pain in Children With Cerebral Palsy Using a Pain Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-0981
Record Dates: First submitted 2009-04-16; First posted 2009-04-21 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Palsy
Keywords: Pain; Pain management; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy; Pain; Agnosia | interventions — Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Analgesic Only (Active Comparator): Group 1 will receive oral analgesic only
  Interventions: Drug: oral analgesic
- anesthetic continuous-infusion + oral analgesia (Active Comparator): Group 2: anesthetic continuous-infusion device, e.g. intravenous analgesic per pump, with supplemental oral analgesia
  Interventions: Drug: intravenous analgesic per pump

INTERVENTIONS:
Drug: oral analgesic — per clinical standard of care
  Arms: Oral Analgesic Only
Drug: intravenous analgesic per pump — per clinical standard of care
  Arms: anesthetic continuous-infusion + oral analgesia

SUMMARY:
The purpose of this study is to determine which pain management strategy continuous analgesic pump or orally-should be used in the management of children with cerebral palsy.

DETAILED DESCRIPTION:
A prospective randomized controlled trial will be performed on up to 150 subjects who will undergo a tendoachilles lengthening, Strayer's procedure, epiphysiodesis of the femur or femoral osteotomy metal work removal.

Subjects will be randomized into two groups: the first group will have an anesthetic pain pump device supplemented with oral analgesia and the second group will only receive oral analgesia. The anesthetic continuous device will be used continuously for 48 hours and with a flow rate of 2ml/hour of 0.25% bupivacaine diluted in accordance to patient weight. Subjects in both groups will receive oral analgesia according to their pain requirements. The amount of oral analgesia used will be documented over 12-hour intervals in a patient diary over a 4 day period. Subjects will have their pain score assessed daily with the use of the Non-Communicating Children's Pain Checklist-Postoperative Version. Their overall satisfaction with post-operative pain management will be assessed at the end of the study with the use of the Parent Total Quality Pain Management questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy between 3 and 17 years old.
* American Society of Anesthesiologists (ASA) intubation grade I, II or III.
* Ability of subject or primary caregivers to give informed consent, to understand what the study entails and to be able to complete the patient Pain Diary during the post-operative period. Subjects should be available for daily telephone follow-up until the data is completed and they should be able to return the completed Pain Diary to the Primary Investigator.
* Willingness and understanding of parent or guardian to have their child randomized to receive either the continuous infusion pain pump device or oral analgesics for their child's pain management.
* English or Spanish-speaking care parent or guardians who are able to complete the Pain Diary.

Exclusion Criteria:

* ASA IV or V,
* Known allergy or sensitivity to bupivacaine,
* Subjects who will have more than the above mentioned procedure performed during their surgical visit,
* Subjects with significant kidney or liver disease,
* Parents/guardians who are assessed by the PI or co-investigators to be unable or unwilling to complete the study's Pain Diary or behavioral tools, and
* Parents/guardians who are unwilling to allow their child to be randomly assigned to receive either the pain pump with oral analgesics or oral medications alone.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2005-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Chang, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- The Children's Hospital, Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Analgesia Only: Group 1 will receive oral analgesia only
- Anesthetic Continuous-Infusion + Oral Analgesia: Group 2 will have an anesthetic continuous-infusion device with supplemental oral analgesia
Period: Overall Study
Arm/Group | Oral Analgesia Only | Anesthetic Continuous-Infusion + Oral Analgesia
Started | 25 | 29
Completed | 16 | 21
Not Completed | 9 | 8
Not completed — Did not return complete pain diaries | 7 | 7
Not completed — Admitted Post-Op | 1 | 0
Not completed — Femoral Stress Fracture | 1 | 0
Not completed — Pain Pump Complication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Group 1 will receive oral analgesia only
- Group 2: Group 2 will have an anesthetic continuous-infusion device with supplemental oral analgesia
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 16 | 21 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 21 | 37
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.1 (2.59) | 8.7 (3.27) | 7.89 (3.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: The Amount of Oral Analgesic Each Subject Consumed Over the 4-day Study Period.
Description: Results of Mean and total Medication administered between the 2 groups over a 4 day period (Mean Medication Administered in mg/kg; SD)
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Oral Analgesia Only | Anesthetic Continuous-Infusion + Oral Analgesia
Number analyzed (Participants) | 16 | 21
mg/kg
  Day 0 | 0.34 (0.26) | 0.24 (0.2)
  Day 1 | 0.39 (0.36) | 0.19 (0.2)
  Day 2 | 0.29 (0.33) | 0.17 (0.19)
  Day 3 | 0.20 (0.27) | 0.09 (0.16)
  Total | 1.22 (1.10) | 0.68 (0.66)

2. Secondary Outcome: Parent and Patient Satisfaction With the Post Operative Pain Management.
Description: Parent responses to questions about pain management traditional paper-based Q method (TPQM) questionnaire.
Time Frame: 4 days
Population: Arms are combined because no outcome measure data is available for separate arms. We have made multiple attempts to contact the PI and study team to obtain data for separate arms. However, the PI has retired and could not be reached, and the study team either could not be reached, has left the university, or did not have the data. Data is only available for 30 parents.
Measure: Count of Participants; unit: Participants
Groups:
- Group I & Group II: Group I: Allocated to receive oral analgesics only Group II: Anesthetic Continuous Infusion + Oral Analgesia
Arm/Group | Group I & Group II
Number analyzed (Participants) | 30
Participants
  Parent felt that pain medicine was able to take away most of their child's pain | 26
  Parent was "Very Satisfied" with child's pain management | 22
  Parent was "Satisfied" with child's pain management. | 7
  Parent was "Dissatisfied" with child's pain management. | 1
  Parent would want their child's pain managed in the same way after another surgery | 28

3. Primary Outcome: The Amount of Pain Analyzed From Pain Scores for Each of the 4 Days.
Description: Pain scores were assessed using a Visual Analog Scale. Possible scores range from 0 (no pain) to 10 (Worst possible pain).
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Analgesia Only | Anesthetic Continuous-Infusion + Oral Analgesia
Number analyzed (Participants) | 16 | 21
score on a scale
  Day 0 | 6.70 (3.21) | 3.79 (2.86)
  Day 1 | 5.17 (2.31) | 2.78 (1.99)
  Day 2 | 3.43 (2.06) | 1.79 (1.44)
  Day 3 | 2.10 (1.68) | 1.74 (2.10)

ADVERSE EVENTS:
Time Frame: 4 days
Groups:
- An Anesthetic Infusion Device With Supplement: Group 2 will have an anesthetic continuous-infusion device with supplemental oral analgesia
Arm/Group | Oral Analgesia Only | An Anesthetic Infusion Device With Supplement
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/21
Other Adverse Events (participants affected / at risk) | 0/16 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No